CLINICAL TRIAL: NCT02900690
Title: Health Economics Evaluation of the Management of Severe Postpartum Hemorrhage: Comparison of Recombinant Activated Factor VII Strategy to the Reference Strategy
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2009/GL
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Health Care Cost; Post Partum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- recombinant activated factor VII (NovoSeven®): Group using the Novoseven
- Standard care: without use of the Novoseven

SUMMARY:
The main objective of this project is to assess the average cost of the treatment of bleeding postpartum with recombinant activated factor VII (NovoSeven®) and compare it to the reference strategy. Costs related to medicine NovoSeven® can generate surplus, but it also avoids in some cases very costly invasive procedures. It will be interesting to compare the average cost of the complete strategies supported.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemorrhage is defined by the following criteria: blood loss greater than 1500 ml graduated measured in the bag and / or hemodynamically unstable and / or requiring transfusion of packed red blood cells (3);
* Sulprostone (Nalador®) ineffective;
* Age over 18 years;
* The term is more than 27 SA (child's viability);
* Without anthropomorphic limit;
* The outcome of the pregnancy is normal or pathological;
* Informed consent "emergency procedure" is signed by the husband or family.

Exclusion Criteria:

* minors, majors in guardianship, with a personal history of venous or arterial thrombosis may cons-indicate treatment with rFVIIa or refuses to sign the consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study is the population described in "rhuFVIIa in Post-partum Hemorrhage " NCT00370877
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2010-11-05 (Actual); Study Completion 2010-11-05 (Actual)

PRIMARY OUTCOMES:
direct medical cost | day 1